CLINICAL TRIAL: NCT06756360
Title: Efficacy and Outcome of Carotid Endarterectomy for Symptomatic Carotid Stenosis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Helal sayed ali, resident doctor at Assiut University hospital, Assiut University
Other Study IDs: carotid endarterectomy
Record Dates: First submitted 2024-12-17; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Carotid Stenosis
Keywords: carotid endarterectomy
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- carotid artery stenosis patient: patients will subjected to Preoperative Carotid doppler - CT angiography Postoperative carotid doppler-CT angiography after 3 days

SUMMARY:
Neurovascular complications can result from this procedure usually from thromboembolism from the operated vessel, cerebral hypoperfusion causing ischaemia and, rarely, intracerebral haemorrhage. The overall incidence of perioperative strokes complicating CEA is approximately 4% ,and represents a devastating outcome that the procedure was designed to prevent. Other neurological sequelae complicating carotid revascularisation include cerebral hyperperfusion syndrome, cranial and peripheral nerve injuries, and contrast encephalopathy in patients undergoing CAS.

The aim of this study is To evaluate the safety and efficacy of carotid endarterectomy for symptomatic carotid Stenosis patients

DETAILED DESCRIPTION:
Carotid stenosis, a condition characterized by the narrowing of the carotid arteries, is a significant concern due to its potential to cause debilitating strokes. As individuals age, the prevalence of moderate to severe carotid artery stenosis increases, particularly after the age of 50, and it affects men more than women. When a physician detects the presence of carotid bruit, an ultrasound examination or CTA/MRA is typically prescribed to confirm the presence and severity of carotid stenosis .

Carotid artery stenosis (CAS) is characterized by the thickening of the arterial walls due to the formation of atherosclerotic plaque, leading to a reduction in the diameter of the artery. The arterial structure is composed of three layers of tissue: tunica intima, tunica media, and tunica adventitia. The tunica intima, which contains a monolayer of endothelial cells, plays a crucial role in facilitating blood movement. In response to injury, the endothelium triggers a biochemical signal for inflammatory cell migration, leading to the formation of fatty streaks and subsequently atherosclerotic plaque. Various factors such as hemodynamic, metabolic, environmental, and genetic risks contribute to inflammatory responses, cell proliferation, and plaque progression. The formation of atheroma in the arterial lumen ultimately results in arterial stenosis, which can lead to transient ischemic attack (TIA) or stroke .

The management of carotid stenosis involves two main interventions: carotid endarterectomy (CEA) and carotid artery stenting (CAS). CEA is a surgical procedure that entails the removal of atherosclerotic material causing stenosis at the carotid bifurcation. It can be performed under local or general anesthesia, with local anesthesia offering the advantage of enabling direct observation and monitoring of the patient's neurological status throughout the procedure. On the other hand, CAS is often carried out under local anesthesia and involves the placement of a stent across the stenosis to restore the normal luminal diameter. Prior to these interventions, patients are typically prescribed lipid-lowering and antithrombotic medications to stabilize the plaque and discourage thrombosis. The indications for CEA and CAS are similar, with considerations for both symptomatic and asymptomatic patients based on the degree of stenosis and the perceived long-term risk of stroke .

. Stroke is prevalent ailment that impacts a substantial number of individuals globally, resulting in both physical impairment and mortality. One of its major causes is carotid artery stenosis. The symptoms and degree of stenosis are key indications for carotid endarterectomy (CEA). In this study, we highlight the indications and outcomes of carotid endarterectomy .

Carotid endarterectomy (CEA) is known to reduce stroke risk in patients with symptomatic, moderate to severe carotid stenosis but has no apparent impact in patients with symptomatic, mild (less than 50%) carotid stenosis. However, recent development of noninvasive imaging modalities has shown that a certain subgroup of patients are at high risk for further ischemic events despite antiplatelet therapy. This study, therefore, aimed to clarify the patients' clinical features and explore the impact of CEA for them.

Carotid artery stenting is an alternative to carotid endarterectomy for the treatment of atherosclerotic carotid artery stenosis.

ELIGIBILITY:
Inclusion Criteria:

* • Symptomatic carotid artery stenosis

  * Carotid artery stenosis more than 60 %

Exclusion Criteria:

* Patient with other etiology (vasculitis dissection)

  * Patient with mild Stenosis
  * Asymptomatic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Symptomatic carotid artery stenosis with Carotid artery stenosis more than 60 %
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
rate of post operative ipsilateral stroke | 30 day
  rate of post operative ipsilateral stroke
mortality rate | 30 day
  short term mortality rate postoperative

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Saxena A, Ng EYK, Lim ST. Imaging modalities to diagnose carotid artery stenosis: progress and prospect. Biomed Eng Online. 2019 May 28;18(1):66. doi: 10.1186/s12938-019-0685-7. PMID 31138235